CLINICAL TRIAL: NCT02108145
Title: Percutaneous Bilateral Versus Unilateral Metal Stent Placement for Hilar Cholangiocarcinoma : A Prospective Open-label Randomized Controlled Trial
Brief Title: Percutaneous Bilateral Versus Unilateral Metal Stent for Hilar Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Head of Department of Digestive Interventional Radiology, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHDD-004
Record Dates: First submitted 2014-03-31; First posted 2014-04-09 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-08

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: cholangiocarcinoma; jaundice; metal stent; PTBS
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma; Jaundice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- unilateral metal stent insertion (Active Comparator): unilateral metal stent insertion was performed either left or right hepatic lobe as can be drainage more liver volume
  Interventions: Procedure: unilateral metal stent insertion
- bilateral metal stent insertion (Experimental): percutaneous transhepatic biliary drainage plus bilateral metal stent.The bare stents were used for PTBS
  Interventions: Procedure: bilateral metal stent insertion

INTERVENTIONS:
Procedure: bilateral metal stent insertion
  Arms: bilateral metal stent insertion
Procedure: unilateral metal stent insertion
  Arms: unilateral metal stent insertion

SUMMARY:
Cholangiocarcinoma (CCA) is the most common biliary malignancy and the second most common hepatic malignancy after hepatocellular carcinoma (HCC). A majority of the CCA (50-70%) was presented in the area of the biliary duct bifurcation. Recent retrospective study included heterogeneous group of malignant diseases demonstrate that draining more than 50% of was associated with a longer median survival.

However, in recent European Society of Gastrointestinal Endoscopy (ESGE) biliary stenting clinical guideline and Asia-Pacific consensus recommendations for endoscopic and interventional management of hilar cholangiocarcinoma (HCCA), whether we should deployment bilateral or unilateral metal stent for patients with HCCA was not clearly recommended due to the absence of randomized controlled trials.

DETAILED DESCRIPTION:
Patients with advanced hilar obstruction (Bismuth III and IV), PTBS had a higher success rate of cholestasis palliation and a low rate of post cholangitis when compared with endoscopic retrograde cholangiopancreatography(ERCP). The advantage of percutaneous approach is the precise lobar selection for drainage and this approach should yield a lower rate of cholangitis.

Guideline recommendation European Society of Gastrointestinal Endoscopy (ESGE) biliary stenting clinical guideline and Asia-Pacific consensus recommendations the goal of palliative stenting of HCCA is drainage of adequate liver volume (50% or more), irrespective of unilateral, bilateral, or multi-segmental stenting was based on heterogeneous group of malignancy by ERCP in retrospective study.There are no randomized clinical trials compared with these two internal biliary drainage methods in HCCA using metal stent.

The aim of the present study was to compare the effect and safety of bilateral versus unilateral stenting in patients with HCCA.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent; Jaundice duo to biliary obstruction; The diagnosis is based on typical features on MRI and magnetic resonance cholangiopancreatography or histologic and cytologic confirmation is established by percutaneous biopsy (X ray-guided) or exploratory laparotomy; Bismuth type Ⅱ、Ⅲ、Ⅳobstruction; Performance status (eastern cooperative oncology group, ECOG) 0-2; All patients were considered unsuitable or refuse for resection on the basis of general medical condition and/or tumor extent.

Exclusion Criteria:

Refuse to participate and provide informed consent; Bismuth Ⅰtype obstruction; Performance status (eastern cooperative oncology group, ECOG) 3-4. Portal Vein involvement; Prior history of stent; Concomitant renal insufficiency; Severe cardiopulmonary diseases; Uncontrolled systemic infection or sepsis; Accompany other malignancy or serious medical illness which may reduce the life expectancy.

Contraindications for PTBS.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-07; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Failure to control jaundice or failure to prevent stent occlusion or re-jaundice within three month after stent implantation | From stent insertion to three months

SECONDARY OUTCOMES:
Median survival | up to 1 year

OTHER OUTCOMES:
Stent patency | up to 1year
  Stent patency is a secondary endpoint of this study. Cumulative stent patency rate is compared between the two groups.
Early major complications | 30 days within treatment
  Early major complications is a secondary endpoint of this study.Early major complications rate is compared between the two groups
30-day mortality | 30 days within treatment
  30-day mortality is a secondary endpoint of this study. 30-day mortality rate is compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, MD,Ph.D, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Han Guo Hong, Xi’an, Shanxi, China